CLINICAL TRIAL: NCT00885443
Title: Emergence Delirium in Children: Total Intravenous Anesthesia With Propofol and Remifentanil Versus Inhalational Sevoflurane Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Carolyne Montgomery, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H08-02470
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-05

CONDITIONS: Emergence Delirium
Keywords: propofol; sevoflurane; pediatric; emergence delirium; Induction of sedation
MeSH Terms: conditions — Emergence Delirium | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Propofol
- 2 (Active Comparator)
  Interventions: Drug: sevoflurane

INTERVENTIONS:
Drug: Propofol — Patients will be anesthetised according to standard induction protocols with propofol/remifentanil intravenously. A laryngeal mask airway (LMA) will be placed by the anesthesiologist, as is usual practice for these cases. A standard dose of fentanyl (1 mcg.kg-1 IV, MAX dose 25 mcg) for postoperative pain and ondansetron (0.1 mg.kg-1 IV, MAX dose 2.5 mg) for PONV prophylaxis will be given to both groups. Dexamethasone will NOT be permitted as an additional antiemetic.
  Arms: 1
Drug: sevoflurane — Patients will be anesthetised according to standard induction protocols with sevoflurane by inhalation. A laryngeal mask airway (LMA) will be placed by the anesthesiologist, as is usual practice for these cases. A standard dose of fentanyl (1 mcg.kg-1 IV, MAX dose 25 mcg) for postoperative pain and ondansetron (0.1 mg.kg-1 IV, MAX dose 2.5 mg) for PONV prophylaxis will be given to both groups. Dexamethasone will NOT be permitted as an additional antiemetic.
  Arms: 2

SUMMARY:
Emergence delirium (ED) refers to a wide variety of behavioural disturbances that are commonly seen in children following emergence from anesthesia. ED can potentially be dangerous and have serious consequences for the child such as injury, increased pain, and dislodgement of medical devices, often requiring physical restraint or pharmacological control. Witnessing this behaviour can be stressful for parents, which can negatively affect their interaction with the healthcare system, and their relationship with the child, nursing staff and other healthcare providers. The investigators aim to minimize ED to reduce the distress experienced by patients and their parents. This study will compare the recovery profile of sevoflurane with that of propofol remifentanil and their associated incidence of ED. This study should enable us to determine which form of anesthesia is associated with the fewest incidences of ED in children.

DETAILED DESCRIPTION:
Purpose:

In children, both propofol-only anesthesia maintenance infusions and single postoperative propofol boluses have been shown to be efficacious at reducing ED when compared with sevoflurane only [13, 17]. Methodological problems in these studies include: the administration of sedative premedications, ED provocative study designs that do not reflect reasonable clinical practice with sevoflurane, and the use of inadequately validated ED outcome tools.

Based on our extensive institutional experience with TIVA, we believe that this technique is superior to sevoflurane with respect to the incidence of ED. However, this clinical impression has never been validated in an appropriately robust investigation, and sevoflurane remains the pediatric anesthetic of choice for most other North American pediatric anesthesiologists.

Hypotheses:

1. The use of total intravenous anesthesia (TIVA), rather than sevoflurane (SEVO) will reduce incidence of ED, as measured by the Pediatric Anesthesia Emergence Delirium (PAED) scale.
2. The use of TIVA will not result in longer times to laryngeal mask airway removal and post anesthetic care unit (PACU) discharge when compared to SEVO.

Objectives:

1. To compare the incidence of ED between SEVO and TIVA anesthesia in children
2. To compare times for recovery from anesthesia between the TIVA and SEVO groups

Research Method:

Recruitment of subjects: With institutional review board approval, and with written informed consent, we will recruit children, ages 2-6 years, undergoing elective strabismus surgery, a relatively minor eye procedure.

Each child will be randomly assigned to one of two groups to receive either TIVA or SEVO. We will exclude children with ASA status IV-V, developmental delay, neurological injury, psychiatric diagnosis, abnormal lipid or carbohydrate metabolism, postoperative nausea or vomiting, Body Mass Index >30, severe anxiety in the pre-operative period requiring sedative premedication or complex medical conditions.

Study design: This study is a randomized, masked clinical trial comparing induction and maintenance of anesthesia with TIVA to SEVO. Every effort will be made to maximize the masking of the observer. All patients will be scored by the Research Fellow, Dr. John Chandler, who will be masked to the anesthetic technique. To evaluate the pre and postoperative state of children we will use of the following scoring tools:

1. The Induction Compliance Checklist (ICC) will be used to evaluate patient preoperative behaviour
2. The PAED scale will be used to assess patients for ED in the PACU.
3. Pain will be assessed postoperatively by means of the face, legs, activity, cry, consolability (FLACC) score currently used in the PACU

Statistical Analysis:

Patients with a PAED score of ≥ 10 will be classified as experiencing ED. Continuous data (weight, BMI) will be analyzed with t-tests and ordinal data (FLACC, PAED, ICC) with Mann-Whitney U tests.

The primary hypothesis will be examined by means of a contingency table and Fisher's exact test.

ELIGIBILITY:
Inclusion Criteria:

* Children having general anesthesia for elective strabismus or other suitable minor eye surgery
* Age ≥ 2 and ≤ 6 years
* ASA I-II
* Appropriate procedure and patient for LMA airway management

Exclusion Criteria:

* Developmental delay or neurological injury
* Psychotropic medications or psychiatric diagnosis
* Abnormal lipid or carbohydrate metabolism
* Deviations from the anesthesia protocol including an inability to secure pre-anesthetic intravenous access in the TIVA group
* Severe anxiety in the pre-operative period requiring sedative. premedication according to the staff anesthesiologist's and family's assessment
* Patients experiencing pain requiring analgesia, postoperative nausea or vomiting (PONV) during the study period
* Patients seen in the pre-anesthetic assessment clinic, due to habituation to hospital environment
* Growth chart percentiles of < 3% or > 97%

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2009-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of emergence delirium | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Carolyne Montgomery, MD, Principal Investigator — University of British Columbia; Mark Ansermino, MD, Study Director — University of British Columbia; Clayton Reichert, MD, Study Director — University of British Columbia; Michelle Misse, Study Chair — British Columbia Children's Hospital; John Chandler, Study Chair — British Columbia Children's Hospital; Disha Mehta, Study Chair — British Columbia Children's Hospital
Locations (1):
- British Columbia Children's Hospital, Vancouver, British Columbia, Canada